CLINICAL TRIAL: NCT00884845
Title: Phase I Multicenter, Open-label, Dose-escalating Clinical and Pharmacokinetic Trial of PM02734 Administered in Combination With Erlotinib in Patients With Advanced Malignant Solid Tumors
Brief Title: Trial of PM02734 Administered in Combination With Erlotinib in Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM2734-A-003-08
Record Dates: First submitted 2009-04-16; First posted 2009-04-21 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: PM2734; Tumors; PharmaMar; Erlotinib; Tarceva
MeSH Terms: conditions — Neoplasms | interventions — elisidepsin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Administration of i.v. infusions of PM02734 (on Days 1, 8 and 15) every three weeks and a daily oral dose of erlotinib
  Interventions: Drug: PM02734 and erlotinib; Drug: Erlotinib

INTERVENTIONS:
Drug: PM02734 and erlotinib — PM02734 drug product (DP) 1 mg/vial is a powder for concentrate for solution for infusion
Drug: Erlotinib — Erlotinib is provided as 25 mg, 100 mg and 150 mg white film-coated tablets
  Other Names: Brand name: TARCEVA

SUMMARY:
Phase I multicenter, open-label, dose-escalating clinical and pharmacokinetic trial of PM02734 administered in combination with erlotinib to determine the safety and tolerability and to identify the dose limiting toxicity (DLT) and the recommended dose (RD) of the combination of PM02734 and erlotinib, in patients with advanced malignant solid tumors.

DETAILED DESCRIPTION:
Phase I multicenter, open-label, dose-escalating clinical and pharmacokinetic trial of PM02734 administered in combination with erlotinib to determine the safety and tolerability and to identify the dose limiting toxicity (DLT) and the recommended dose (RD) of the combination of PM02734 and erlotinib, determine the preliminary pharmacokinetics (PK) of the combination, evaluate the preliminary PK/pharmacodynamic correlation, evaluate the preliminary antitumor activity, perform a preliminary pharmacogenomic (PGx) study to explore molecular predictors of response to ErbB receptor antagonists and PM02734 in patient with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent form.
* Histologically or cytologically confirmed advanced malignant solid tumors.
* Measurable or non-measurable disease following (RECIST)
* Age ≥ 18 years.
* Life expectancy ≥ 3 months.
* Performance status ECOG ≤ 2.
* Recovery from any drug-related adverse events (AEs) derived from previous treatments.
* Appropriate bone marrow, liver and renal function.
* Left ventricular ejection fraction (LVEF) within normal limits for the institution.
* Women of childbearing potential must have a negative serum pregnancy test before study entry. Both men and women must agree to use a medically acceptable method of contraception throughout the treatment period and for three months after discontinuation of treatment.

Exclusion Criteria:

* Prior therapy with PM02734.
* Pregnant or lactating women.
* Less than four weeks from radiation therapy.
* Evidence of progressive central nervous system (CNS) metastases. or any symptomatic brain or leptomeningeal metastases.
* Other relevant diseases or adverse clinical conditions.
* Any other major illness that, in the Investigator's judgment.
* Limitation of the patient's ability to comply with the treatment or to follow-up at a participating protocol.
* Ingestion of potent cytochrome CYP3A4 inhibitors.
* Treatment with any investigational product in the 30-day period prior to the first infusion.
* Known hypersensitivity to any component of PM02734 or erlotinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability and to identify the dose limiting toxicity (DLT) and the recommended dose (RD) of the combination of PM02734 and erlotinib | 2 years

SECONDARY OUTCOMES:
To determine preliminary: pharmacokinetics (PK) , PK / pharmacodynamic correlation, antitumor activity, pharmacogenomic (PGx) study to explore molecular predictors of response. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Roman Pérez-Soler, M.D., Principal Investigator — Montefiore Medical Center (NY - USA); Rafael Rosell, M.D., Principal Investigator — Hospital Universitario Germans Trias i Pujol (Badalona - Spain); Mauricio Cuello, M.D., Principal Investigator — Instituto Universitario Dexeus (Barcelona - Spain)
Locations (3):
- Montefiore Medical Center, New York, New York, United States
- Spain (2):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Intituto Universitario Dexeus, Barcelona, Barcelona